CLINICAL TRIAL: NCT06986928
Title: A Network Analysis on the Role of Specific Emotion Regulation Abilities as Emotional Resilience Factors for Distress and Mental Health, in Relation to Childhood Abuse Exposure in Adolescents and Young Adults
Brief Title: A Network Analysis on the Role of Specific ER Abilities as ERFs for Distress and Mental Health, in Relation to CAs Exposure in the AYAs
Status: Completed | Type: Observational
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor PhD, Babes-Bolyai University
Other Study IDs: REThinkRESILIENT-Network
Record Dates: First submitted 2025-04-24; First posted 2025-05-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Emotional Resilience

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents and young adults: Adolescents and young adults will be recruited from various schools and university programs in Cluj-Napoca.
  Interventions: Other: No intervention will be applied.

INTERVENTIONS:
Other: No intervention will be applied. — No intervention will be applied.
Other: No intervention will be applied. — No intervention will be implemented in this study, as the questionnaires will serve an exploratory purpose.

SUMMARY:
This activity will aim to compare the network of emotional resilience factors and stress in adolescents and young adults depending on the childhood abuse exposure (considered moderator), using a network analysis approach.

DETAILED DESCRIPTION:
Participants included in this study (age range = 10-24, G*power estimated N = 349) will complete a set of questionnaires on constructs that are focusing on or closely related to resilience and mental health, in order to investigate the dynamics of emotional resilience factors in relation to mental health outcomes such as anxiety and depression, taking into account the moderating effects of childhood abuse exposure.

ELIGIBILITY:
Inclusion Criteria:

* adolescents and young adults between 10 and 24 years old provided with written parental consent where applicable

Exclusion Criteria:

* intellectual disability or physical limitations precluded the use of the computer program

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: School- and university-aged students recruited from educational institutions in Cluj-Napoca.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Childhood Trauma Exposure | Baseline
  Childhood Trauma Screener (CTS)
Emotion regulation abilities | Baseline
  The REThink Life game-based emotion regulation abilities will be assessed using a scenario of social exclusion and measuring the use of using different emotion regulation strategies.
Emotional and behavioral difficulties | Baseline
  Strengths and Difficulties Questionnaire (SDQ)
Stress | Baseline
  Adolescence Stress Scale (ADOSS)

CONTACTS AND LOCATIONS:
Overall Officials: Oana A. David, Ph.D, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No